CLINICAL TRIAL: NCT03744221
Title: Health Effects of Sustainable Future Proteins
Acronym: Su-Pro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Diederik Esser, project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL65835.081.18
Record Dates: First submitted 2018-11-02; First posted 2018-11-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-11

CONDITIONS: Intestinal Barrier Function; Protein Digestion Kinetics

STUDY DESIGN:
Intervention Model Description: double blind, randomised, cross-over, short-term trial in which 36 study subject will participate. Study subjects will receive three protein interventions of 1 week with a washout period of 1 week between interventions. 12 subjects will also receive an acute postprandial digestibility test at the start of the intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Proteins will be packed in non-transparent sealed sachets/jars and labeled with 'protein A/B/C'. Proteins will be flavored to mask taste
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Corn protein (Experimental): Corn protein powder
  Interventions: Dietary Supplement: Corn protein powder
- Bovine plasma protein (Experimental): Bovine plasma protein powder
  Interventions: Dietary Supplement: Bovine plasma protein powder
- control benchmark protein Whey (Active Comparator): Whey protein powder
  Interventions: Dietary Supplement: Whey protein powder

INTERVENTIONS:
Dietary Supplement: Corn protein powder — 40g/d ( 2 times 20 grams per day for a period of 1 week)
  Other Names: sustainable protein source 1
  Arms: Corn protein
Dietary Supplement: Bovine plasma protein powder — 40g/d ( 2 times 20 grams per day for a period of 1 week)
  Other Names: sustainable protein source 2
  Arms: Bovine plasma protein
Dietary Supplement: Whey protein powder — 40g/d ( 2 times 20 grams per day for a period of 1 week)
  Other Names: control protein source
  Arms: control benchmark protein Whey

SUMMARY:
In the current study the investigators aim to assess the nutritional quality and bio-functional activity of two alternative protein sources bovine plasma and corn and from the benchmark protein whey. The study is a double blind, randomised, cross-over, short-term trial in which 36 healthy study subjects will receive three protein interventions of 1 week with a washout period of 1 week between interventions. Study subjects will visit the research facility before and after the intervention period on two separate occasions to measure gut permeability via a multi-sugar test and to collect fasting blood samples and blood pressure outcomes. Faecal and saliva samples before and after each intervention will be collected. A subgroup of 12 study participants will also be subjected to a postprandial digestibility test on the first day of the interventions. The main study parameter is to assess the protein digestion kinetics and protection of the epithelial barrier. Secondary study parameters include other markers of gastrointestinal health, metabolic health, vascular health and satiating properties.

DETAILED DESCRIPTION:
In the current study the investigators aim to assess the nutritional quality and bio-functional activity of two alternative protein sources bovine plasma and corn and from the benchmark protein whey. The objective is to assess the degree of digestibility and protection of the epithelial barrier of two alternative protein concentrates from corn and bovine plasma and of the commonly consumed benchmark protein whey. These outcomes will also be used to evaluate how predictive the in vitro-measurements have been for the obtained in vivo-effects. Secondary objectives are to assess the impact on other markers of gastrointestinal health, metabolic health, vascular health and satiating properties. Study design: The study is a double blind, randomised, cross-over, short-term trial in which 36 study subject will participate. Study subjects will receive three protein interventions of 1 week with a washout period of 1 week between interventions. Study subjects will visit the research facility before and after the intervention period on two separate occasions to measure gut permeability via a multi-sugar/acetylsalicylic acid test and to collect fasting blood samples and blood pressure outcomes. Faecal and saliva samples before and after each intervention will be collected. All measurements will be conducted after an overnight fast and a standardised evening meal prior to the study days. A subgroup of 12 study participants will also be subjected to a postprandial digestibility test on the first day of the interventions.

Study population: healthy study subjects, between 35-70y, BMI 18 - 30kg/m2, both males and females.

Intervention (if applicable): Three intervention arms of one week; a bovine plasma protein intervention, a corn protein intervention and a whey protein comparator intervention. Study subjects will receive 40 grams of protein per day during the intervention in two 20 g doses.

Main study parameters/endpoints: The main study parameter is to assess the protein digestion kinetics and protection of the epithelial barrier. Secondary study parameters include other markers of gastrointestinal health, metabolic health, vascular health and satiating properties.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Age between 35-70 y
* BMI between 18 - 30 kg/m2

Exclusion Criteria:

* Intake of medications known to change the inflammatory status (including proton pump inhibitors, anti-inflammatory medication (including NSAIDs)
* Having a history of medical or surgical events that may significantly affect the study outcome
* Kidney dysfunction (self-reported)
* Gastrointestinal disorders, constipation (defecation <3 times a week) or history of gastrointestinal surgery
* Allergies for our intervention products
* Recent use of antibiotics (<1 month prior to day 01 of the study)
* Not having a general practitioner
* Mental status that is incompatible with the proper conduct of the study
* Pregnancy or lactating
* Reported weight loss or weight gain of > 5 kg in the month prior to pre-study screening
* Reported slimming, medically prescribed, other (extreme) diet, or use of protein concentrates
* Not willing to give up blood donation during the study
* Current smokers
* Alcohol intake > 3 glasses per day
* Hard-drug abuse
* Participation in other clinical trials in the past month
* Being an employee or student of the department Consumer Science & Health group of Wageningen Food & Biobased Research

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Change in gut permeability for total cohort | before (Day-1) and after (Day6) the protein intervention
  multi-sugar acetylsalicylic acid test
Change in blood free amino acids (e.g. Degree of digestibility) on a subset of participants | before (Day0) each intervention, 20 gram protein will be consumed and blood samples will be taken before and up to 3 hours after protein consumption
  postprandial test, determine free amino acids in blood samples collected before and after the postprandial challenge test

SECONDARY OUTCOMES:
change in blood markers of intestinal health, | before (Day0) and after (Day7) the protein intervention, under fasting conditions
  like diamine oxidase, A1AT, citrulline, FABP-2, CRP or complement,
change in faecal microbiota | before (Day0) and after (Day7) the protein intervention
  obtained from fecal samples
change in faecal metabolites | before (Day0) and after (Day7) the protein intervention
  obtained from faecal samples
change in VAS scores on intestinal complains | daily during the intervention from day1 until day7 of the intervention
  On a scale ranging from worst-best outcome (higher scores are better)

OTHER OUTCOMES:
change in blood pressure | before (Day0) and after (Day7) the protein intervention, under fasting conditions
  Systolic and diastolic blood pressure
change in Pulse Wave Analysis | before (Day0) and after (Day7) the protein intervention, under fasting conditions
  augmentation index
change in Glucose | before (Day0) and after (Day7) the protein intervention, under fasting conditions and after postprandial protein intake
  Blood markers of metabolic health
change in Insulin | before (Day0) and after (Day7) the protein intervention, under fasting conditions and after postprandial protein intake
  Blood markers of metabolic health
change in saliva markers | before (day-1 and day0) and after (day6 and day7) the protein intervention
  reflecting intestinal health

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Esser, Dr, Principal Investigator — Wageningen research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
will not be shared